CLINICAL TRIAL: NCT06214130
Title: Multiple-dose, Randomized, Open-Label, Fasting, Two-period, Crossover, Bioavailability Study Between Orfiril Long 500 mg Prolonged-Release Minitablets and Ergenyl Chrono 500 mg Prolonged-Release Tablets in Healthy, Male Volunteers.
Brief Title: Bioavailability of Orfiril Long 500 mg Prolonged-Release Minitablets and Ergenyl Chrono 500 mg Prolonged-Release Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Desitin Arzneimittel GmbH (Industry)
Collaborators: BioPharma Services Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VPA-056/K
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Multiple Drug Use
MeSH Terms: interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Orfiril long 500 mg (sodium valproate) prolonged-release minitablets
  Interventions: Drug: Sodium valproate 500 MG; Drug: Valproic Acid 500 MG
- Reference (Active Comparator): Ergenyl chrono 500 mg (valproic acid) prolonged -release tablets
  Interventions: Drug: Sodium valproate 500 MG; Drug: Valproic Acid 500 MG

INTERVENTIONS:
Drug: Sodium valproate 500 MG — oral intake
  Other Names: Orfiril long 500 mg
Drug: Valproic Acid 500 MG — oral intake
  Other Names: Ergenyl chrono 500 mg

SUMMARY:
Comparative bioavailability of valproate from Orfiril long 500 mg prolonged-release mini-tablets and Ergenyl chrono 500 mg prolonged-release tablets in healthy, male volunteers under fasting conditions.

DETAILED DESCRIPTION:
Pivotal, multiple-dose, randomized, open-label, two-period, two-sequence, two-treatment, single-centre, crossover, study designed to evaluate the comparative bioavailability of valproate for Orfiril long 500 mg prolonged release minitablets and Ergenyl chrono 500 mg prolonged-release tablet once daily for 6 days in healthy male subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking (from at least 6 months prior to study drug administration), male volunteers, 18-65 years of age, inclusive.
2. BMI that was between 18.5 and 30.0 kg/m², inclusive.
3. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
4. Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, and heart rate between 50-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
5. Clinical laboratory values within BPSI's most recent acceptable laboratory test range, and/or values were deemed by the PI/Sub-Investigator as "Not Clinically Significant".
6. Ability to comprehend and be informed of the nature of the study, as assessed by BPSI staff. Capable of giving written informed consent prior to any study- related procedure. Must have been to communicate effectively with clinic staff.
7. Ability to fast for at least 14 hours and consume standard meals.
8. Availability to volunteer for the entire study duration and was to adhere to all protocol requirements.
9. Agreed not to have a tattoo or body piercing until the end of the study.
10. Agreed not to receive the COVID-19 vaccination from 7 days prior to the first study drug dose until 7 days after the last study drug administration in the study.
11. Agreed not to drive or operate heavy machinery if feeling dizzy or drowsy following study drug administration until full mental alertness was regained.
12. Males who were able to father children must agree to use medically acceptable methods of contraception and to not donate sperm during the study and for 60 days after the last study drug administration.

Medically acceptable methods of contraception include using a condom with a female partner of child-bearing potential who was using oral contraceptives, hormonal patch, implant or injection, intrauterine device, or diaphragm with spermicide. Abstinence as a method of contraception is acceptable if it was in line with the preferred and usual lifestyle of the study participant.

If a subject's partner became pregnant during his participation in the study and for 60 days after he has completed his last study drug administration, he must have informed BPSI staff immediately.

Exclusion Criteria:

Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.

2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first study drug administration, as determined by the PI/Sub-Investigator.

3. Estimated creatinine clearance <70 ml/min. 4. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.

5. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.

6. A positive test result for any of the following: HIV, Hepatitis B surface antigen, Hepatitis C, drugs of abuse (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), breath alcohol test and cotinine.

7. Known history or presence of:

* Alcohol abuse or dependence within one year prior to first study drug administration;
* Drug abuse or dependence;
* Hypersensitivity or idiosyncratic reaction to Orfiril Long, its excipients, and/or related substances;
* Suicidal ideation or suicidal behavior, as assessed by the Columbia Suicide Severity Rating Scale (baseline version) - Appendix B (Refer to Appendix 16.1.1)
* Food allergies;
* Presence of any dietary restrictions unless deemed by the PI/Sub-I as "Not Clinically Significant".
* Family history of hereditary neurometabolic syndromes due to mitochondrial enzyme polymerase;
* Family history of liver disease;
* Known urea cycle disorder;
* Known porphyria;
* Coagulation disorder;
* Severe allergic reactions (e.g., anaphylactic reactions, angioedema). 8. Intolerance to and/or difficulty with blood sampling through venipuncture. 9. Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets etc.

  10. Individuals who have donated, in the days prior to first study drug administration:
* 50-499 mL of blood in the previous 30 days;
* 500 mL or more in the previous 56 days. 11. Donated plasma by plasmapheresis within 7 days prior to first study drug administration.

  12. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first study drug administration.

  13. Use of any enzyme-modifying drugs and/or other products, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., barbiturates, carbamazepine, glucocorticoids, phenytoin, St. John´s Wort, and rifampicin) in the previous 30 days before first study drug administration.

  14. Used of any monoamine oxidase (MAO) inhibitors (e.g., phenelzine, tranylcypromine) within 30 days prior to first study drug administration.

  15. Used of any prescription medication within 14 days prior to first study drug administration.

  16. Used of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements) within 14 days prior to first study drug administration.

  17. Consumed food or beverages containing grapefruit and/or pomelo within 10 days prior to first study drug administration.

  18. Consumed food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing in each study period.

  19. Individuals who had undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.

  20. Difficulty with swallowing whole tablets. 21. Unable or unwilling to provide informed consent. 22. Had a tattoo or body piercing within 30 days prior to first study drug administration.

  23. A subject who, in the opinion of the investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Area under the curve during steady state (AUCtau, ss) | Day 6: pre-dose (0), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 18 and 24 hours post-dose.
  Comparative bioavailability under fasting steady state conditions, the 90% confidence intervals (CI) for the Test/Reference ratios of geometric means for AUCtau,ss should fall within 80.00%-125.00%.
Maximal plasma concentration during steady state (Cmaxss) | Day 6: pre-dose (0), 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 18 and 24 hours post-dose.
  Comparative bioavailability under fasting steady state conditions, the 90% confidence intervals (CI) for the Test/Reference ratios of geometric means for AUCtau,ss should fall within 80.00%-125.00%.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Faulknor, MD, Principal Investigator — BioPharma Services Inc.
Locations (1):
- Biopharma Services INC, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No